CLINICAL TRIAL: NCT07143175
Title: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation (CARE-D-Foot-Nav), a Single-arm Pilot Study
Brief Title: CARE-D-FOOT-Nav Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Marcos C. Schechter, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008869
Record Dates: First submitted 2025-08-08; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Foot Ulcer (DFU)
Keywords: Assistance for Effective Diabetic Foot Navigation; Navigators; Wound care; Wound healing
MeSH Terms: conditions — Diabetic Foot | interventions — Health Resources

STUDY DESIGN:
Intervention Model Description: Single-arm prospective study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will be assigned a dedicated DFU patient navigator.
  Interventions: Other: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation

INTERVENTIONS:
Other: Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation — The CARE-D-FOOT-Nav (Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation) program is a patient navigator intervention that aims to increase access to guideline-concordant multidisciplinary DFU care to improve DFU healing.
  CARE-D-Foot-Nav is a diabetes educator who will serve as a dedicated Diabetic Foot Ulcer (DFU) patient navigator. The navigator will assist the subjects with diabetic foot ulcer care.
  Based on community input, navigators will conduct 30-to 60-minute encounters, either by phone or in person, at least once a week during the 20-week program. Additional contact may be warranted to coordinate appointments and transportation. Participants can call the navigator with DFU-related concerns at any time during the navigator's working hours. The overarching goal of the navigator is to help patients access the four key pillars of DFU care, thereby optimizing the chances of DFU healing.
  Other Names: CARE-D-Foot-Nav; Diabetic Foot Navigator

SUMMARY:
This pilot study aims to examine the implementation of a patient navigator intervention called Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation (CARE-D-Foot-Nav).

Up to one-third of the 37 million people living with diabetes in the United States will experience a diabetic foot ulcer in their lifetime, and non-healing diabetic foot ulcers are the reason for almost all 100,000 diabetes-related amputations that occur annually in this country. Multidisciplinary diabetic foot care improves ulcer healing; however, people face challenges in navigating the healthcare system to access high-quality, multidisciplinary care, and amputations are on the rise.

Participants enrolled in Care-D-Foot-Nav will be assigned to a diabetes educator and/or registered dietitian, and/or medical assistant who will serve as a dedicated DFU patient navigator. The navigators will conduct 30-60-minute encounters by phone or in person at least once a week during the 20-week program. The navigator will provide additional resources depending on the unique needs and circumstances of the participant. In addition, participants may receive transportation assistance and wound care supplies if needed.

This pilot study aims to evaluate the program's fidelity and acceptability. The findings of this study may provide a new and cost-effective approach to managing this devastating disease.

DETAILED DESCRIPTION:
The CARE-D-Foot-Nav (Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation) study is a pilot trial testing whether a patient navigator-led intervention can improve healing outcomes for patients hospitalized with diabetic foot ulcers (DFUs). DFUs are a serious complication of diabetes that contribute to over 100,000 amputations annually in the U.S. and account for a significant portion of diabetes-related healthcare costs. DFU healing rates remain low in the US. DFUs that fail to heal within 30 days are at a higher risk. Unfortunately, there is a resurgence in diabetes-related amputations. Healing requires complex, multidisciplinary care, focused on glycemic control, wound management, vascular disease treatment, and infection therapy. A strategy to facilitate multidisciplinary DFU care and support patients in their healing journey that can be widely implemented is essential to improve DFU healing rates and curb the diabetes-related limb loss pandemic, particularly for underserved and high-risk populations.

Patient navigators are healthcare personnel who mitigate barriers to care by facilitating care logistics, connecting patients to available resources, and promoting patient engagement. While navigators have been shown to improve diabetes outcomes, their effectiveness in improving DFU care and promoting healing remains untested. Informed by extensive preliminary data and community input, the investigators developed the CARE-D-Foot-Nav (Comprehensive Assistance and Resources for Effective Diabetic Foot Navigation) program.

This study aims to determine whether the CARE-D-Foot-Nav program improves DFU healing rates, enhances patient engagement, and can be implemented cost-effectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old) with diabetes admitted to the hospital for any reason who undergo a DFU-related amputation of 2 or more digits (including minor and major amputations)
* English-speaking patients (available patient navigators are English-speaking).

Exclusion Criteria:

* Patients who are unable to understand the nature and scope of the study,
* Enrolled in another clinical trial,
* Planned discharge to an acute or long-term care facility,
* Planning to receive outpatient DFU care outside of Grady.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of the program components addressed | Up to 20 weeks during program participation
  Researchers will measure the program fidelity by the proportion of the program components addressed by the navigators. Navigators will address 16 components during the weekly encounters and 22 components at every fourth encounter. Researchers will record all encounters and will listen to the recordings of encounters and count which components were or were not discussed (binary outcome, yes/no), and measure consistency across navigators.
Acceptability of the CARE-D-Foot-Nav intervention | Up to 20 weeks during program participation
  Researchers will conduct focus group discussions and/or one-on-one interviews with the participants to understand the program's likes and dislikes. There is no measuring scale.

SECONDARY OUTCOMES:
Number of participants with wound healing with complete re-epithelialization of the wound. | Baseline and week 20 (day 140 +/- 7 days)
  Researchers will measure the effectiveness of the intervention by the wound healing. Researchers will take pictures of the wounds at enrollment and week 20 (day 140 +/- 7 days), and two independent reviewers who are clinical DFU experts, will review the pictures to ascertain wound healing. To minimize the missing data, participants who miss the final 20-week visit will be asked to send pictures of their feet. If >1 DFU is present, wound healing assessment will be based on the largest wound. If participants experience amputation or death before week 20, the ulcer will be classified as not healed.
Number of participants with confirmed wound healing | Baseline and week 22
  Researchers will measure the effectiveness of the intervention based on wound healing. Photographs of the wounds will be taken at enrollment and again at week 22 (i.e., approximately two weeks ±7 days after the participant's primary outcome visit). Two independent reviewers, who are clinical DFU experts, will evaluate the photographs to determine whether wound healing has occurred.
  If more than one DFU is present, the assessment will be based on the largest wound. If a participant undergoes an amputation or dies before week 20, the ulcer will be classified as not healed.
DFU care clinic attendance | At 14 days and 30 days after hospital discharge
  DFU care clinic attendance within 14- and 30-days of hospital discharge, defined as attending outpatient visits with any provider managing a) diabetes, b) wound care, c) antibiotics for DFU infection, if applicable, and (d) obtaining non-invasive PAD testing if not done in the last 12 months. Researchers will measure these outcomes singly and in combination.
Wound area reduction | Baseline and week 20
  Difference in diabetic foot ulcer areas will be reported.
Major amputations | After hospital discharge (up to 20 weeks)
  Number of subjects undergoing amputation above the ankle.
Number of amputations | After hospital discharge (up to 20 weeks)
  Number of subjects undergoing any type of amputation (major or minor) after hospital discharge.
Mortality | After hospital discharge (up to 20 weeks)
  Number of deaths after hospital discharge during the study period.
Change in hemoglobin A1c | Baseline and week 20
  Researchers will measure glycemic control by the change in hemoglobin A1c.
EuroQol five-dimensional (EQ-5D) score | Baseline and week 20
  The EuroQol 5-Dimension (EQ-5D) is a standardized instrument used to measure health-related quality of life. It's a self-report questionnaire that assesses health across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a few levels of severity, allowing individuals to describe their health state. Each dimension has five levels: 1 = no problems, to 5 = extreme problems/unable to do. The five answers produce a unique 5-digit health state, for example, 11234, that describes the young person's health state. For example, the code 11234 describes a health state where there are no problems with walking about (mobility) or looking after myself, a little bit of a problem with doing usual activities, some pain or discomfort, and feeling really worried, sad, or unhappy.
Diabetic foot ulcer - short form (DFS-SF) score | Baseline and week 20
  A short form of the Diabetic Foot Ulcer Scale (DFS) is called the Diabetic Foot Ulcer Scale-Short Form (DFS-SF). It's a 29-item questionnaire designed to assess the impact of diabetic foot ulcers on a patient's quality of life (QOL), grouped into six subscales: leisure, physical health, dependence/daily life, negative emotions, worried about ulcers/feet, and bothered by ulcer care. Each item is scored on a 5-point Likert scale, ranging from 1 = "not at all" to 5 = "very common". Each subscale is scored on a scale of 0 to 100. Higher scores on the DFS-SF indicate a better quality of life, while lower scores indicate a poorer quality of life.
  The minimum score for each subscale is 0, representing the worst QOL, and the maximum score is 100, representing the best QOL.
Change in the Interpersonal Support Evaluation List-12 | Baseline and week 20
  Perceived social support will be measured using the Interpersonal Support Evaluation List-12. The Interpersonal Support Evaluation List-12 (ISEL-12) is a brief, validated questionnaire designed to assess perceived availability of social support. The ISEL-12 includes 12 items that evaluate the perceived support across three dimensions: Appraisal Support, Belonging Support, and Tangible Support.
  Each item is rated on a 4-point Likert scale. Scores range from 12 to 48, with higher scores indicating greater perceived social support and low scores indicating lower social support.
Change in the Trust in Physicians' Scale | Baseline and week 20
  Medical mistrust will be measured using the Trust in Physicians Scale. Trust in Physicians Scale is used to measure interpersonal trust a patient has in their individual physician.
  Each item is rated on a 5-point Likert scale. Total score range: 11 (low trust) to 55 (high trust).
  Higher scores indicate greater trust in the physician.
Tobacco cessation | Baseline and 20 weeks
  Self-reported cessation at week 20 among those reporting tobacco use at baseline.
Acute care utilization | up to 20 weeks after hospital discharge
  All-cause emergency department (ED) visits and re-hospitalizations after hospital discharge.
Services accessed | Baseline and 20 weeks
  Services accessed (e.g., foodbank) after hospital discharge ascertained through electronic medical record review and participant interviews.
Food insecurity | Baseline and 20 weeks
  Food insecurity will be assessed via validated EHR-embedded survey items. Food insecurity severity is often assessed based on the number of affirmative responses. More affirmative responses typically indicate greater food insecurity.
Housing stability | Baseline and 20 weeks
  Housing Stability will be assessed using survey items embedded in the electronic health record (EHR). Responses are coded as:
  0 = Stable housing (e.g., own/rent a steady place to live)
  1 = Unstable housing (e.g., temporarily staying with others, in a shelter, or without a place to live)
  Scores will be summarized as the proportion of participants with unstable housing at baseline and week 20.
Financial resource strain questionnaire | Baseline and 20 weeks
  Financial resource strain scoring assesses the level of difficulty individuals experience in meeting their basic living expenses and financial obligations, assessed via validated EHR-embedded survey items. A score of 27 on the Financial Strain Questionnaire indicates greater financial strain than a score of 9. Lower scores/categories indicate less financial strain. Higher scores indicate greater strain
Transportation needs | Baseline and 20 weeks
  Transportation needs will be assessed via a validated EHR-embedded transportation survey from the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experiences (PRAPARE) tool.
  The transportation tool is a 2-question survey where "yes" indicates transportation needs. More affirmative responses typically indicate increased transportation needs.
Peer support group attendance | After hospital discharge (up to 20 weeks)
  Proportion of CARE-D-Foot-Nav participants who attended ≥1 peer support group meetings and number of meetings attended.

OTHER OUTCOMES:
Costs and resource utilization | After hospital discharge (up to 20 weeks)
  Total resource utilization cost per participant over the study period will be calculated by converting the following components to standardized U.S. dollar equivalents and summing time navigators spend with participants and coordinating care, time providers spend discussing participant care with navigators, number of outpatient visits scheduled by navigators, and the cost of wound care supplies, phones dispensed, and transportation.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Schechter, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia

IPD SHARING:
Plan to Share IPD: No